CLINICAL TRIAL: NCT05189496
Title: Study on the Effectiveness and Safety of Hyperbaric Oxygen Therapy for Preventing Radiation Pneumonitis Caused by Radiotherapy and Chemotherapy of Breast Cancer
Brief Title: Hyperbaric Oxygen in the Prevention of Radiation Pneumonitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KY-Q-2021-182
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Radiation Pneumonitis
Keywords: Hyperbaric Oxygen; Radiation Pneumonitis; Breast Cancer; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Radiation Pneumonitis; Breast Neoplasms | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyperbaric oxygen therapy group (Experimental): 30-40 times hyperbaric oxygen therapy
  Interventions: Behavioral: hyperbaric oxygen therapy
- control group (No Intervention): No hyperbaric oxygen therapy

INTERVENTIONS:
Behavioral: hyperbaric oxygen therapy — hyperbaric oxygen therapy
  Arms: hyperbaric oxygen therapy group

SUMMARY:
Radiotherapy is one of the important treatments to improve the survival rate of breast cancer patients, but also has the risk of radiation lung injury, which can develop into pulmonary fibrosis. Hyperbaric oxygen can improve the tissue after radiation by promoting the function of vascular endothelial cells and fibroblasts, and reducing the secretion of inflammatory factors, thereby inhibiting the process of fibrosis and fiber atrophy after radiotherapy, and promoting tissue repair. Therefore, it has the potential value of treating chronic radiation injury. We aim to investigate whether hyperbaric oxygen treatment can reduce the incidence of radiation pneumonia and improve patients' quality of life, and to evaluate its safety and the impact on the patients' long-term survival outcomes.

DETAILED DESCRIPTION:
Radiotherapy is one of the important treatments to improve the survival rate of breast cancer patients. Radiotherapy also has the risk of radiation lung injury, which can develop into pulmonary fibrosis, which seriously affects the quality of life of patients. Hyperbaric oxygen has received more attention in the field of delayed tissue damage caused by radiotherapy. In a hyperbaric oxygen environment, sufficient oxygen supply can improve the tissue after radiation by promoting the function of vascular endothelial cells and fibroblasts, and reducing the secretion of inflammatory factors. Low blood vessel density, low cell activity and low oxygen content in the "three low" state, thereby inhibiting the process of fibrosis and fiber atrophy after radiotherapy, and promoting tissue repair. Therefore, it has the potential value of treating chronic radiation injury. Can hyperbaric oxygen therapy be applied for breast cancer patients who were receiving radiotherapy, reduce the risk of radiation pneumonitis, prevent radiation pneumonitis and even radiofibrosis, and improve long-term survival? Therefore, we plan to prospectively enroll 380 breast cancer patients and randomly divide them into two groups. The treatment group will be given 30-40 hyperbaric oxygen therapy immediately after the end of radiotherapy, to study whether hyperbaric oxygen therapy reduces the risk of radiation pneumonia, and to evaluate hyperbaric oxygen The safety of treatment and its impact on the patient's quality of life and long-term survival outcomes provide an effective means to reduce the incidence of radiation pneumonia and improve the long-term quality of life.

ELIGIBILITY:
Inclusion Criteria:

* (1) Volunteer to participate and sign informed consent in writing. (2) Past pathological diagnosis of breast cancer followed by radical treatment/surgery for breast cancer, followed by adjuvant chemotherapy followed by radiotherapy.

  (3) Excluding patients with simple neck lymph node recurrence and patients with distant metastases.

  (4) There is no secondary malignant tumor in other parts. (5) Age at entry ≥ 18 years old and ≤ 70 years old, both male and female. (6) The Eastern Cooperative Oncology Group (ECOG) has a performance status score of 0 or 1.

  (7) The expected survival period is ≥2 years. (8) There was no acute radiation lung injury in chest CT examination before and after radiotherapy

Exclusion Criteria:

* (1) Contraindications to hyperbaric oxygen therapy: lung disease (severe chronic obstructive airway disease, bullous lung disease, acute or chronic lung infection, uncontrolled asthma, untreated pneumothorax), in the past History of ear surgery, middle ear disease (eustachian tube dysfunction, recurrent dizziness), eye disease (retinal detachment).

  (2) Have received hyperbaric oxygen therapy in the past. (3) Radiation pneumonia had occurred at the time of enrollment or before receiving hyperbaric oxygen therapy.

  (4) Women who are pregnant or breastfeeding. (5) Patients who have not completed comprehensive breast cancer treatment due to disease progression, intolerable side effects, abandonment of treatment and other reasons.

  (8) Patients who need mechanical ventilation support. (9) Patients who cannot follow and understand simple commands. (10) Patients with disorientation and mental disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiation pneumonitis | 1 year
  Rate of enrolled participants with radiation pneumonitis

SECONDARY OUTCOMES:
Grade of symptoms related to radiation pneumonitis | 1 year
  The severity of symptoms (cough, shortness of breath, and so on) related to radiation pneumonitis, which is based on the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grading scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.